CLINICAL TRIAL: NCT01107054
Title: A Double Blind, Randomized, Multiple Dose, Placebo And Active Controlled 4-Way Crossover Study To Investigate The Effects Of Inhaled PF-00610355 On QT/QTC Interval In Healthy Subjects
Brief Title: A Study to Investigate the Effects of PF00610335 on the QT/QTC Interval in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A7881014
Record Dates: First submitted 2010-04-19; First posted 2010-04-20 (Estimated); Last update posted 2011-01-13 (Estimated); Status verified 2011-01

CONDITIONS: Pulmonary Disease; Lung Disease; Moxifloxacin
Keywords: QTC
MeSH Terms: conditions — Lung Diseases | interventions — N-((4'-hydroxybiphenyl-3-yl)methyl)-2-(3-(2-((-2-hydroxy-2-(4-hydroxy-3-((methylsulfonyl)amino)phenyl)ethyl)amino)-2-methylpropyl)phenyl)acetamide; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- PF-00610355 450 µg (Experimental): An orally inhaled dose of PF-00610355 450 µg
  Interventions: Drug: PF-00610355
- PF-00610355 1200 µg (Experimental): An orally inhaled dose of PF-00610355 1200 µg
  Interventions: Drug: PF-00610355
- moxifloxacin 400 mg (Active Comparator): A single oral dose of moxifloxacin 400 mg on Day 4.
  Interventions: Drug: moxifloxacin
- placebo (Placebo Comparator): A single oral dose of non-matched placebo on Day 4.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: PF-00610355 — An orally inhaled dose of PF-00610355 450 µg on days 1 to 4
  Arms: PF-00610355 450 µg
Drug: PF-00610355 — An orally inhaled dose of PF-00610355 1200 µg on days 1 to 4
  Arms: PF-00610355 1200 µg
Drug: moxifloxacin — A single oral dose of moxifloxacin 400 mg on Day 4.
  Arms: moxifloxacin 400 mg
Drug: placebo — A single oral dose of non-matched placebo on Day 4.
  Arms: placebo

SUMMARY:
A study to determine the cardiovascular effects of PF00610335 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects aged 18 to 55 years
* Informed consent document signed by the subject or a legally acceptable representative
* Subjects who are willing and able to comply with the scheduled visits, treatment tests, laboratory tests, and other study procedures

Exclusion Criteria:

* Evidence or history of clinically significant haematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic psychiatric, neurologic or allergic disease or clinical findings at screening
* Conditions possibly affecting drug absorption
* 12-lead ECg demonstrating QTc > 450ms or any other clinically significant abnormalities at screen
* Positive urine drug screen
* Hypersensitivity to moxifloxacin or PF00610335
* Unwilling or unable to comply with the lifestyle guidelines in the protocol Treatment with an investigational drug within 3 months or 5 half lives (whichever is longer) preceding the first dose of study medication

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2010-06; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To assess whether multiple dose administration of PF00610335 has the potential to affect QTc in healthy volunteers | 24 hours

SECONDARY OUTCOMES:
To assess the effects of a positive control (moxifloxacin) on QTc interval in healthy volunteers | 24 hours
To asses the the relationship between plasma concentrations of PF00610335 and its effects, if any on the QTc interval | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7881014&StudyName=A%20Study%20to%20investigate%20the%20effects%20of%20PF00610335%20on%20the%20QT/QTC%20interval%20in%20healthy%20volunteers